CLINICAL TRIAL: NCT06486415
Title: Serial Measurement of Beta-Human Chorionic Gonadotropin (BHCG) Values During the Day in the Diagnosis of Ectopic Pregnancy
Brief Title: Novel Diagnosis of Ectopic Pregnancy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Acibadem Ob&Gyn
Record Dates: First submitted 2024-06-06; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Ectopic Pregnancy; hCG; Pregnancy of Unknown Location
Keywords: ectopic pregnancy; hCG; Pregnancy with unknown location
MeSH Terms: conditions — Pregnancy, Ectopic

STUDY DESIGN:
Intervention Model Description: In participants with clinically suspected ectopic pregnancy who come to the Gynecology clinic with menstrual delay and high Beta Human Chorionic Gonadotropin (BHCG) levels, serum BHCG values will be checked 5 times with 2-hour intervals on the same day. 10 ectopic pregnancy and 10 normal pregnancy patients will be included in the study. The serum BHCG increase trend of patients whose normal pregnancy was clinically detected by ultrasound despite the suspicion of ectopic pregnancy, and the change trend in serum BHCG of patients whose diagnosis of ectopic pregnancy is confirmed will be analyzed and compared. Diagnostic criteria for BHCG change in ectopic pregnancy will be established according to the differences in the serum BHCG increase trend.
  This is an interventional study. Taking 5 blood samples of the ectopic pregnancy patients in the same day are the interventions of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ectopic pregnancy patients (Experimental): the group diagnosed as ectopic pregnancy after serial testing of Beta Human Chorionic Gonadotropin (BHCG) levels
  Interventions: Diagnostic Test: serum BHCG testing
- Normal pregnancy (Active Comparator): The group diagnosed with normal pregnancy after serial measurements of serum BHCG levels.
  Interventions: Diagnostic Test: serum BHCG testing

INTERVENTIONS:
Diagnostic Test: serum BHCG testing — Taking 5ml blood samples every 2 hours for 5 times for measurement of BHCG. Blood samples will be taken from the median cubital and cephalic veins which is located inner side of the elbow.

SUMMARY:
In the project, the investigators aim to determine the Beta- human chorionic gonadotropin (BHCG) value with serial measurements on the same day in the diagnosis of ectopic pregnancy.

DETAILED DESCRIPTION:
Ectopic pregnancy is when the conception material is in a location other than the endometrial cavity. The diagnosis of ectopic pregnancy is basically made by the lack of increase in serum BHCG values as in normal pregnancy. In normal pregnancies, BHCG value increases by 70% or more every 2 days. In ectopic pregnancy, an increase of less than 70% every 2 days is diagnostic. This classical method allows the diagnosis to be made within 2-4 days at the earliest. Most of the time, this period can take 6-10 days.

In the project, the investigators will investigate how to determine the BHCG value with serial measurements on the same day in the diagnosis of ectopic pregnancy. The fact that there is no 70% increase after 2 days in ectopic pregnancy suggests that there may be an irregular increase during the day. The investigators aim to make this diagnosis in a shorter time than long days by measuring BHCG values many times during the day in patients with suspected ectopic pregnancy. The fact that there is no other study on this subject in the literature strengthens the possibility of the project being published as valuable information for the literature, even if a negative result is obtained as a result of this study.

ELIGIBILITY:
Inclusion Criteria:

* Positive bhcg levels

Exclusion Criteria:

* clinically diagnosis of intrauterine pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Beta-hCG Levels Measured Every 2 Hours as a Discriminating Factor Between Ectopic and Normal Pregnancy | 10 hours
  The primary outcome is how the changes in Beta-hCG levels measured every two hours differ between the ectopic pregnancy and the normal pregnancy.

SECONDARY OUTCOMES:
Increase pattern of BHCG levels in normal pregnancy | 10 hours
  BHCG increase pattern every two hours in normal pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Ozguc Takmaz, Assoc.Prof., Principal Investigator — Acibadem Maslak Hospital

IPD SHARING:
Plan to Share IPD: Yes
If requested, data will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available after submission of the trail results to a scientific journal.
Access Criteria: Data will be shared in a publicly accessible web site.